CLINICAL TRIAL: NCT02680574
Title: Phase 3, Randomized, Open-label, Active-controlled Study Evaluating the Efficacy and Safety of Oral Vadadustat for the Maintenance Treatment of Anemia in Subjects With Non-dialysis-dependent Chronic Kidney Disease (NDD-CKD) (PRO2TECT-CONVERSION)
Brief Title: Efficacy and Safety Study to Evaluate Vadadustat for the Maintenance Treatment of Anemia in Participants With Non-dialysis-dependent Chronic Kidney Disease (NDD-CKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0015; 2015-004774-14 (EudraCT Number)
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Results first posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Anemia; Non-Dialysis-Dependent Chronic Kidney Disease
Keywords: Vadadustat; AKB-6548; Chronic kidney disease; anemia; CKD; chronic renal insufficiency; renal impairment; erythropoietin; kidney; renal; oral anemia treatment; hemoglobin; hypoxia-inducible factor; HIF; hypoxia-inducible factor prolyl-hydroxylase inhibitor; HIF-PHI; efficacy; safety; Phase 3; cardiovascular; NDD-CKD
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — vadadustat; Darbepoetin alfa

STUDY DESIGN:
Masking Description: Sponsor was blinded during the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vadadustat (Experimental)
  Interventions: Drug: Vadadustat
- Darbepoetin alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Vadadustat — Oral dose administered once daily for ≥36 weeks. Dose adjustment based on hemoglobin level as defined in the protocol.
  Other Names: AKB-6548
  Arms: Vadadustat
Drug: Darbepoetin alfa — Subcutaneous or intravenous dose administered for ≥36 weeks. Initial dose based on the current package insert for investigational sites in the United States (US), and the Summary of Product Characteristics for all other investigational sites (non-US) for adult participants with chronic kidney disease not on dialysis. For participants already on Darbepoetin alfa, the initial dosing regimen in the study was based on the prior dosing regimen.
  Other Names: Aranesp
  Arms: Darbepoetin alfa

SUMMARY:
A multicenter, randomized, open-label, active-controlled Phase 3 study for the maintenance treatment of anemia in participants with Non-dialysis-dependent Chronic Kidney Disease (NDD-CKD)

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, active-controlled Phase 3 study of the efficacy and safety of Vadadustat versus Darbepoetin alfa for the maintenance treatment of anemia in participants with NDD-CKD

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Diagnosis of chronic kidney disease (CKD) with an estimated glomerular filtration rate ≤60 milliliters per minute per 1.73 square meter (mL/min/1.73 m^2) at Screening and not expected to start dialysis within 6 months of Screening
* Currently maintained on erythropoiesis-stimulating agents therapy, with a dose received within 6 weeks prior to or during Screening
* Mean Screening hemoglobin between 8.0 and 11.0 grams per deciliter (g/dL) (inclusive) in the United States (US) and between 9.0 and 12.0 g/dL (inclusive) outside of the US
* Serum ferritin ≥100 nanograms per milliliter (ng/mL) and transferrin saturation (TSAT) ≥20% during Screening

Exclusion Criteria:

* Anemia due to a cause other than CKD or participant with active bleeding or recent blood loss
* Red blood cell transfusion within 8 weeks prior to randomization
* Uncontrolled hypertension
* Severe heart failure at Screening (New York Heart Association Class IV)
* Acute coronary syndrome (hospitalization for unstable angina or myocardial infarction), surgical or percutaneous intervention for coronary, cerebrovascular, or peripheral artery disease (aortic or lower extremity), surgical or percutaneous valvular replacement or repair, sustained ventricular tachycardia, hospitalization for heart failure, or stroke within 12 weeks prior to or during Screening
* Hypersensitivity to Darbepoetin or Vadadustat or to any of their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1725 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (404):
- United States (184):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Tuscumbia, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Anaheim, California
  - Research Site, Bakersfield, California
  - Research Site #1, Chula Vista, California
  - Research Site #2, Chula Vista, California
  - Research Site, El Centro, California
  - Research Site, Fountain Valley, California
  - Research Site, Glendale, California
  - Research Site, Granada Hills, California
  - Research Site, La Mesa, California
  - Research Site, Laguna Hills, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site #1, Northridge, California
  - Research Site #2, Northridge, California
  - Research Site, Riverside, California
  - Research Site, Roseville, California
  - Research Site, Salinas, California
  - Research Site, San Diego, California
  - Research Site #1, San Dimas, California
  - Research Site #2, San Dimas, California
  - Research Site, Santa Ana, California
  - Research Site, Santa Monica, California
  - Research Site, Sherman Oaks, California
  - Research Site, Thousand Oaks, California
  - Research Site, Whittier, California
  - Research Site, Arvada, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Westminster, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Bradenton, Florida
  - Research Site, Brandon, Florida
  - Research Site, Cooper City, Florida
  - Research Site #1, Coral Gables, Florida
  - Research Site #2, Coral Gables, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Doral, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Hialeah, Florida
  - Research Site #1, Hialeah, Florida
  - Research Site #2, Hialeah, Florida
  - Research Site #3, Hialeah, Florida
  - Research Site #1, Hollywood, Florida
  - Research Site #2, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site #1, Jacksonville, Florida
  - Research Site #2, Jacksonville, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site #1, Miami, Florida
  - Research Site #2, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site #1, Miami Lakes, Florida
  - Research Site #2, Miami Lakes, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site #1, Columbus, Georgia
  - Research Site #2, Columbus, Georgia
  - Research Site #1, Lawrenceville, Georgia
  - Research Site #2, Lawrenceville, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, McHenry, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Jeffersonville, Indiana
  - Research Site #1, Merrillville, Indiana
  - Research Site #2, Merrillville, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Monroe, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Greenbelt, Maryland
  - Research Site, Takoma Park, Maryland
  - Research Site, Methuen, Massachusetts
  - Research Site, Plymouth, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Port Huron, Michigan
  - Research Site, Roseville, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Gulfport, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Butte, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site #1, Las Vegas, Nevada
  - Research Site #2, Las Vegas, Nevada
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Berlin, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Santa Fe, New Mexico
  - Research Site, Flushing, New York
  - Research Site, Laurelton, New York
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site #1, Greenville, North Carolina
  - Research Site #2, Greenville, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Jersey Shore, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Sumter, South Carolina
  - Research Site, West Columbia, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Dallas, Texas
  - Research Site, DeSoto, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Gonzales, Texas
  - Research Site, Greenville, Texas
  - Research Site, Houston, Texas
  - Research Site #1, Houston, Texas
  - Research Site #2, Houston, Texas
  - Research Site, Lewisville, Texas
  - Research Site #1, McAllen, Texas
  - Research Site #2, McAllen, Texas
  - Research Site, McKinney, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sherman, Texas
  - Research Site, Victoria, Texas
  - Research Site, Clinton, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, St. George, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Alexandria, Virginia
  - Research Site, Arlington, Virginia
  - Research Site, Danville, Virginia
  - Research Site, Hampton, Virginia
  - Research Site, Lansdowne Town Center, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Salem, Virginia
  - Research Site, Woodbridge, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Wenatchee, Washington
  - Research Site, Madison, Wisconsin
- Argentina (17):
  - Research Site, Bahía Blanca, Buenos Aires
  - Research Site, Junín, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Pergamino, Buenos Aires
  - Research Site, Ramos Mejía, Buenos Aires
  - Research Site, San Miguel, Buenos Aires
  - Research Site, San Nicolás de los Arroyos, Buenos Aires
  - Research Site, Sarandí, Buenos Aires
  - Research Site, Temperley, Buenos Aires
  - Research Site, Godoy Cruz, Mendoza Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Salta
  - Research Site, San Luis
- Australia (12):
  - Research Site, Camperdown, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Cairns, Queensland
  - Research Site, Gold Coast, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Launceston, Tasmania
  - Research Site, Bentleigh East, Victoria
  - Research Site, Box Hill, Victoria
  - Research Site, Fitzroy, Victoria
  - Research Site, Nedlands, Western Australia
  - Research Site, Perth, Western Australia
- Austria (2):
  - Research Site, Sankt Pölten
  - Research Site, Vienna
- Brazil (21):
  - Research Site, Fortaleza, Ceará
  - Research Site, Vitória, Espírito Santo
  - Research Site, Feira de Santana, Estado de Bahia
  - Research Site, Itabuna, Estado de Bahia
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Juiz de Fora, Minas Gerais
  - Research Site, Curitiba, Paraná
  - Research Site #1, Curitiba, Paraná
  - Research Site #2, Curitiba, Paraná
  - Research Site, Maringá, Paraná
  - Research Site, Rio de Janeiro, Rio Do Janeiro
  - Research Site, Caxias do Sul, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Criciúma, Santa Catarina
  - Research Site, Joinville, Santa Catarina
  - Research Site, Botucatu, São Paulo
  - Research Site, Campinas, São Paulo
  - Research Site, Santo André, São Paulo
  - Research Site, São Bernardo do Campo, São Paulo
  - Research Site, São Paulo, São Paulo
- Bulgaria (13):
  - Research Site, Byala
  - Research Site, Cherven Bryag
  - Research Site, Lom
  - Research Site, Silistra
  - Research Site, Sliven
  - Research Site, Smolyan
  - Research Site, Sofia
  - Research Site #1, Sofia
  - Research Site #2, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Vratsa
- Research Site, Scarborough Village, Ontario, Canada
- Chile (4):
  - Research Site, Concepción
  - Research Site, Puerto Varas
  - Research Site, Santiago
  - Research Site, Temuco
- Colombia (7):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Espinal
  - Research Site, Manizales
  - Research Site #1, Medellín
  - Research Site #2, Medellín
  - Research Site, Medellín
- Czechia (3):
  - Research Site, České Budějovice
  - Research Site, Hradec Králové
  - Research Site, Prague
- France (6):
  - Research Site, Lille, Alpes De Haute Provence
  - Research Site, Reims, Marne
  - Research Site, Saint-Priest-En-Jarez, Pays de la Loire Region
  - Research Site, Pontoise, Val d'Oise
  - Research Site, Créteil, Val De Marne
  - Research Site, Paris
- Germany (5):
  - Research Site, Villingen-Schwenningen, Baden-Wurttemberg
  - Research Site, Rostock, Mecklenburg-Vorpommern
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Berlin
  - Research Site, Hamburg
- Hungary (14):
  - Research Site #1, Baja
  - Research Site #2, Baja
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Esztergom
  - Research Site, Hódmezővásárhely
  - Research Site, Kalocsa
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Kistarcsa
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Szigetvár
- Israel (5):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Nahariya
  - Research Site, Ramat Gan
  - Research Site, Rishon LeZiyyon
- Italy (11):
  - Research Site, Piedimonte Matese, Caserta
  - Research Site, San Giovanni Rotondo, Foggia
  - Research Site, Bari
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site #1, Napoli
  - Research Site #2, Napoli
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Siena
- Malaysia (3):
  - Research Site, Alor Star, Kedah
  - Research Site, Kuala Lumpur
  - Research Site, Pulau Pinang
- Mexico (15):
  - Research Site, Torreón, Coahuila
  - Research Site, Acapulco de Juárez, Guerrero
  - Research Site #1, Pachuca, Hidalgo
  - Research Site #2, Pachuca, Hidalgo
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Morelia, Michoacán
  - Research Site, Monterrey, Nuevo León
  - Research Site, San Juan del Río, Querétaro
  - Research Site, Culiacán, Sinaloa
  - Research Site, Mazatlán, Sinaloa
  - Research Site, Chihuahua City
  - Research Site, Durango
  - Research Site, Veracruz
- New Zealand (2):
  - Research Site, Hamilton
  - Research Site, New Plymouth
- Research Site, Nowa Sól, Poland
- Research Site, Caguas, Puerto Rico
- Romania (5):
  - Research Site, Bucharest
  - Research Site #1, Bucharest
  - Research Site #2, Bucharest
  - Research Site, Oradea
  - Research Site, Timișoara
- Russia (9):
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Krasnoyarsk
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Petrozavodsk
  - Research Site, Pushkin
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Serbia (7):
  - Research Site #1, Belgrade
  - Research Site #2, Belgrade
  - Research Site #3, Belgrade
  - Research Site, Kragujevac
  - Research Site, Lazarevac
  - Research Site, Niš
  - Research Site, Zaječar
- Slovakia (5):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Galanta
  - Research Site, Svidník
  - Research Site, Trstená
- South Africa (9):
  - Research Site, Bloemfontein, Free State
  - Research Site, Winnie Mandela, Free State
  - Research Site, Pretoria, Gauteng
  - Research Site, Vereeniging, Gauteng
  - Research Site #1, Durban, KwaZulu-Natal
  - Research Site #2, Durban, KwaZulu-Natal
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Tongaat, KwaZulu-Natal
  - Research Site, Worcester, Western Cape
- South Korea (7):
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Guri-si, Gyeonggi-do
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seoul
- Spain (12):
  - Research Site, Elche, Alicante
  - Research Site, Torrevieja, Alicante
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, L'Hospitalet de Llobregat, Barcelona
  - Research Site, Málaga, Málaga
  - Research Site, Almería
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Seville
  - Research Site, Valencia
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Erciyes
  - Research Site, Istanbul
  - Research Site, Kocaeli
- Ukraine (11):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kropyvnytskyi
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Mykolaiv
  - Research Site, Odesa
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
- United Kingdom (8):
  - Research Site, Exeter, Devon
  - Research Site, London, Greater London
  - Research Site, Salford, Greater Manchester
  - Research Site, Stevenage, Hertfordshire
  - Research Site, Leicester, Leicestershire
  - Research Site, Kings Lynn, Norfolk
  - Research Site, Doncaster, South Yorkshire
  - Research Site, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chertow GM, Eckardt KU, Sarnak MJ, Winkelmayer WC, Agarwal R, Minga T, Luo W, Burke SK. Safety and Efficacy of Vadadustat for the Treatment of CKD-Related Anemia within and outside the United States. J Am Soc Nephrol. 2025 Oct 1;36(10):1984-1997. doi: 10.1681/ASN.0000000708. Epub 2025 May 13. PMID 40359056
- [Derived] Parfrey PS, Burke SK, Chertow GM, Eckardt KU, Jardine AG, Lewis EF, Luo W, Matsushita K, McCullough PA, Minga T, Winkelmayer WC. Safety Endpoints With Vadadustat Versus Darbepoetin Alfa in Patients With Non-Dialysis-Dependent CKD: A Post Hoc Regional Analysis of the PRO2TECT Randomized Clinical Trial of ESA-Treated Patients. Kidney Med. 2023 May 12;5(7):100667. doi: 10.1016/j.xkme.2023.100667. eCollection 2023 Jul. PMID 37427292
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Chertow GM, Pergola PE, Farag YMK, Agarwal R, Arnold S, Bako G, Block GA, Burke S, Castillo FP, Jardine AG, Khawaja Z, Koury MJ, Lewis EF, Lin T, Luo W, Maroni BJ, Matsushita K, McCullough PA, Parfrey PS, Roy-Chaudhury P, Sarnak MJ, Sharma A, Spinowitz B, Tseng C, Tumlin J, Vargo DL, Walters KA, Winkelmayer WC, Wittes J, Eckardt KU; PRO2TECT Study Group. Vadadustat in Patients with Anemia and Non-Dialysis-Dependent CKD. N Engl J Med. 2021 Apr 29;384(17):1589-1600. doi: 10.1056/NEJMoa2035938. PMID 33913637

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2961 participants were screened for entry into the study. Of these, 1725 participants were enrolled and randomized into the study.
Groups:
- Vadadustat: Participants were randomized to receive Vadadustat at an initial oral dose of 300 milligrams per day (mg/day). Thereafter, Vadadustat was taken once daily on an outpatient basis. Up-and-down titration to 150, 300, 450, and 600 mg (available tablet strength was administered as the appropriate number of 150 mg tablets) was allowed during the study based on hemoglobin (Hb) level measurements to maintain target Hb levels.
- Darbepoetin Alfa: Participants were randomized to Darbepoetin alfa at an initial dose that was based on the current package insert for investigational sites in the United States (US), and the Summary of Product Characteristics (SmPC) for all other investigational sites (non-US) for adult participants with chronic kidney disease not on dialysis. For participants already on Darbepoetin alfa, the initial dosing regimen in the study was based on the prior dosing regimen.
Period: Overall Study
Arm/Group | Vadadustat | Darbepoetin Alfa
Started | 862 | 863
Completed | 704 | 711
Not Completed | 158 | 152
Not completed — Death | 137 | 137
Not completed — Withdrawal by Subject | 17 | 9
Not completed — Lost to Follow-up | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vadadustat | Darbepoetin Alfa | Total
Number analyzed (Participants) | 862 | 863 | 1725
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (13.14) | 66.5 (13.52) | 66.9 (13.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 468 | 488 | 956
  Male | 394 | 375 | 769
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 32 | 26 | 58
  Asian | 62 | 55 | 117
  Black or African American | 93 | 131 | 224
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  White | 631 | 603 | 1234
  Not Reported | 15 | 13 | 28
  Reported as Other | 25 | 32 | 57
  Multiple | 1 | 3 | 4
Average hemoglobin [Mean (Standard Deviation); unit: Grams per deciliter (g/dL)] | 10.423 (0.8871) | 10.390 (0.9430) | 10.406 (0.9154)
Mean estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 22.6 (11.64) | 22.8 (12.04) | 22.7 (11.84)
Number of Participants with History of Diabetes [Count of Participants; unit: Participants] | 444 | 432 | 876
Number of Participants with NYHA Functional Classification of Heart Failure [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) functional classification serves as a fundamental descriptor of heart failure. NYHA heart failure classes are as follows: Class 0 (no congestive heart failure [CHF]), Class I (No symptoms and no limitation in ordinary physical activity), Class II (Mild symptoms and slight limitation during ordinary activity), Class III (Marked limitation in activity due to symptoms, even during less-than-ordinary activity), and Class IV (Severe limitations. Experiences symptoms even while at rest). NYHA class IV is also an exclusion criteria.
  Participants
    NYHA Class 0 | 610 | 595 | 1205
    NYHA Class I | 108 | 108 | 216
    NYHA Class II | 113 | 122 | 235
    NYHA Class III | 29 | 36 | 65
    NYHA Class IV | 0 | 0 | 0
    NYHA Class Missing | 2 | 2 | 4
Number of Participants with Any History of Heart Failure [Count of Participants; unit: Participants]
  Yes | 44 | 52 | 96
  No | 613 | 595 | 1208
  Missing | 205 | 216 | 421

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin (Hb) to the Average Over the Primary Efficacy Period (Weeks 24 to 36)
Description: The Baseline average was calculated as the average of the Hb values obtained at the screening visit closest to the date of randomization and the randomization visit. The average for the Primary Efficacy Period was calculated as the average Hb value over Weeks 24 to 36. Analysis was conducted using an analysis of covariance (ANCOVA) model with multiple imputation for missing data with Baseline hemoglobin concentration (<10.0 versus ≥10.0 g/dL), geographic region (United States [US] versus European Union [EU] versus Rest of World [ROW]), and New York Heart Association congestive heart failure (NYHA CHF) class (Class 0 [no CHF] or I versus II or III) as covariates.
Time Frame: Baseline; Weeks 24 to 36
Population: Randomized Population: All participants randomized. Analyses of this population were based on the randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter (g/dL)
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 862 | 863
Grams per deciliter (g/dL) | 0.41 (0.036) | 0.42 (0.037)
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Treatment comparison: Vadadustat minus Darbepoetin Alfa; Test type: Non-Inferiority — Establishment of non-inferiority was based on a margin of -0.75 g/dL applied to the difference in mean change of hemoglobin: Vadadustat minus Darbepoetin alfa; Least squares mean difference = -0.01, 95% CI 2-sided [-0.09 to 0.07], Standard Error of Mean 0.042

2. Primary Outcome: Median Time to First Major Adverse Cardiovascular Event (MACE)
Description: MACE was defined as all-cause mortality, non-fatal myocardial infarction (MI), or non-fatal stroke. The primary safety outcome was positively adjudicated first MACE, which was defined as any death, Endpoint Adjudication Committee (EAC)-confirmed non-fatal MI, or EAC-confirmed non-fatal stroke occurring between the first dose date and each participant's last participation date. PROTECT MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Results and statistical analysis from study AKB-6548-CI-0015 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0014 and AKB-6548-CI-0015 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to Week 208
Population: Safety Population (PRO2TECT): All participants from the PRO2TECT (Non-dialysis-dependent chronic kidney disease [NDD-CKD]) population who received 1 or more doses of study drug. Only those participants with MACE events were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 168 | 152
Weeks | 53.21 [30.64 to 81.43] | 58.00 [31.07 to 99.21]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0015 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per Food and Drug Administration [FDA]) and 1.3 (per European Medicines Agency [EMA]); p = 0.2015, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.930 to 1.446]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Time to first MACE for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 382 and 344 respectively; median time to first event (Q1, Q3) = 50.07 (23.00, 82.86) weeks versus 51.93 (27.79, 91.00) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.0725, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [1.012 to 1.355]

3. Secondary Outcome: Change From Baseline in Hb to the Average Over the Secondary Efficacy Period (Weeks 40 to 52)
Description: The Baseline average was calculated as the average of the Hb values obtained at the screening visit closest to the date of randomization and the randomization visit. The average for the Secondary Efficacy Period was calculated as the average Hb value over Weeks 40 to 52. Analysis was conducted using an ANCOVA model with multiple imputation for missing data with Baseline hemoglobin concentration (<10.0 versus ≥10.0 g/dL), geographic region (US versus EU versus ROW), and NYHA CHF class (Class 0 [no CHF] or I versus II or III) as covariates.
Time Frame: Baseline; Weeks 40 to 52
Population: Randomized Population. Analyses of this population were based on the randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 862 | 863
g/dL | 0.43 (0.044) | 0.44 (0.044)
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Treatment comparison: Vadadustat minus Darbepoetin Alfa; Test type: Non-Inferiority — Establishment of non-inferiority was based on a margin of -0.75 g/dL applied to the difference in mean change: Vadadustat minus Darbepoetin alfa; Least squares mean difference = -0.00, 95% CI 2-sided [-0.10 to 0.09], Standard Error of Mean 0.05

4. Secondary Outcome: Median Time to First MACE Plus Hospitalization for Heart Failure or Thromboembolic Event Excluding Vascular Access Thrombosis
Description: MACE was defined as all-cause mortality, non-fatal MI, or non-fatal stroke. Hospitalization for EAC adjudicated heart failure included presentation of participants to an acute care facility requiring an overnight hospitalization (change in calendar day) with an exacerbation of heart failure requiring treatment. EAC confirmed thromboembolic events for this secondary outcome measure included arterial thrombosis, deep vein thrombosis, and pulmonary embolism. PROTECT MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Results and statistical analysis from study AKB-6548-CI-0015 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0014 and AKB-6548-CI-0015 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to Week 208
Population: Safety Population (PRO2TECT). Only those participants with MACE plus hospitalization for heart failure or thromboembolic event excluding vascular access thrombosis were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 197 | 195
Weeks | 48.29 [22.71 to 72.71] | 49.29 [20.14 to 86.43]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0015 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.7770, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.851 to 1.268]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Time to first MACE plus hospitalization for heart failure or thromboembolic events excluding vascular access thrombosis for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 451 and 424 respectively; median time to first event (Q1, Q3) = 42.86 (19.71, 73.43) weeks versus 43.86 (21.36, 80.43) weeks, respectively; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.2305, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.972 to 1.267]

5. Secondary Outcome: Median Time to First Cardiovascular MACE
Description: MACE was defined as all-cause mortality, non-fatal MI, or non-fatal stroke. Cardiovascular MACE analysis differed from the primary MACE endpoint as it included only deaths adjudicated by the EAC as cardiovascular deaths (i.e, only EAC-confirmed cardiovascular deaths) in addition to first events of non-fatal MI or non-fatal stroke. PROTECT MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Results and statistical analysis from study AKB-6548-CI-0015 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0014 and AKB-6548-CI-0015 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to Week 208
Population: Safety Population (PRO2TECT). Only those participants with cardiovascular MACE events were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 89 | 83
Weeks | 45.57 [20.14 to 67.57] | 50.29 [18.29 to 83.29]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0015 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.5509, Gray's Test; Based on non-parametric analysis; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.817 to 1.501]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Time to first cardiovascular MACE for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 198 and 178 respectively; median time to first event (Q1, Q3) = 45.57 (21.71, 73.29) weeks versus 47.36 (20.00, 88.43) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.2531, Gray's Test; Based on non-parametric analysis; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.947 to 1.420]

6. Secondary Outcome: Median Time to First Cardiovascular Death
Description: Cardiovascular death included EAC adjudicated fatal MI, pump failure, sudden death, presumed sudden death, fatal stroke, fatal pulmonary embolism, cardiovascular procedure-related death, other cardiovascular death, and presumed cardiovascular death. PROTECT MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Results and statistical analysis from study AKB-6548-CI-0015 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0014 and AKB-6548-CI-0015 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to Week 208
Population: Safety Population (PRO2TECT). Only those participants with cardiovascular death were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 56 | 66
Weeks | 48.29 [29.50 to 69.14] | 54.21 [30.71 to 94.14]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0015 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.4184, Gray's test; Based on non-parametric analysis; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.610 to 1.258]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Time to first cardiovascular death for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 127 and 131 respectively; median time to first event (Q1, Q3) = 48.29 (28.86, 76.14) weeks versus 48.43 (21.29, 92.29) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.8613, Gray's test; Based on non-parametric analysis; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.792 to 1.293]

7. Secondary Outcome: Median Time to First All-cause Mortality
Description: Only events that were positively adjudicated and confirmed by the EAC were included in the MACE analyses. PROTECT MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Results and statistical analysis from study AKB-6548-CI-0015 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0014 and AKB-6548-CI-0015 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to Week 208
Population: Safety Population (PRO2TECT). Only those participants with all-cause mortality were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 139 | 139
Weeks | 57.71 [35.29 to 87.00] | 62.14 [34.14 to 111.57]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0015 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.8041, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.820 to 1.315]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Time to first all-cause mortality for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 319 and 307 respectively; median time to first event (Q1, Q3) = 52.14 (28.71, 84.71) weeks versus 53.00 (30.71, 94.14) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.4577, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.930 to 1.274]

8. Other Pre Specified Outcome: Exploratory - Proportion of Participants With Hb Values Within the Target Range During the Primary Evaluation Period (Weeks 24 to 36)
Time Frame: Weeks 24 to 36
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Exploratory - Proportion of Time With Hb Values Within the Target Range During the Primary Evaluation Period (Weeks 24 to 36)
Time Frame: Weeks 24 to 36
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory - Proportion of Time With Hb Values Within the Target Range During the Secondary Evaluation Period (Weeks 40 to 52)
Time Frame: Weeks 40 to 52
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Exploratory - Proportion of Participants With Hb Values Within the Target Range During the Secondary Evaluation Period (Weeks 40 to 52)
Time Frame: Weeks 40 to 52
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Exploratory - Proportion of Participants With an Hb Increase of >1.0 g/dL From Baseline Visit
Time Frame: Baseline; up to Week 52
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Exploratory - Time to Achieve Hb Increase of >1.0 g/dL From Baseline Visit
Time Frame: Baseline; up to Week 52
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Exploratory - Mean Change in Hb Between Baseline (Mean Pretreatment Hb) and the Primary Evaluation Period (Mean Hb From Weeks 24 to 36) Stratified by Pre-baseline Erythropoiesis-stimulating Agent (ESA) Exposure
Time Frame: Baseline; Weeks 24 to 36
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Exploratory - Mean Monthly Dose of Intravenous (IV) Elemental Iron Administered in Participants Who Have Received IV Iron
Time Frame: Up to Week 52
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Exploratory - Proportion of Participants Receiving IV Iron Therapy
Time Frame: Up to Week 52
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Exploratory - Proportion of Participants Receiving Red Blood Cells (RBCs) Transfusion(s)
Time Frame: Up to Week 52
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 208 weeks
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began (or pre-existing AEs that worsened) on or after the first dose through each participant's last participation date, were reported in study AKB-6548-CI-0015 (NCT02680574). Of the participants randomized, 1723 participants were included in the Safety population (861 and 862 participants in the Vadadustat and Darbepoetin alfa treatment groups, respectively). Two randomized participants did not receive treatment.
Arm/Group | Vadadustat | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 139/861 | 139/862
Serious Adverse Events (participants affected / at risk) | 504/861 | 488/862
Other Adverse Events (participants affected / at risk) | 482/861 | 436/862
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat (N=861) | Darbepoetin Alfa (N=862)
End stage renal disease (Renal and urinary disorders) | 232 | 238
Pneumonia (Infections and infestations) | 56 | 49
Acute kidney injury (Renal and urinary disorders) | 34 | 32
Cardiac failure congestive (Cardiac disorders) | 29 | 31
Acute myocardial infarction (Cardiac disorders) | 34 | 24
Urinary tract infection (Infections and infestations) | 20 | 20
Anaemia (Blood and lymphatic system disorders) | 16 | 18
Death (General disorders) | 20 | 13
Sepsis (Infections and infestations) | 17 | 16
Cardiac failure acute (Cardiac disorders) | 15 | 16
Atrial fibrillation (Cardiac disorders) | 16 | 13
Cardiac failure (Cardiac disorders) | 10 | 19
Fluid overload (Metabolism and nutrition disorders) | 17 | 12
Dehydration (Metabolism and nutrition disorders) | 16 | 10
Cardiac arrest (Cardiac disorders) | 9 | 16
Cellulitis (Infections and infestations) | 6 | 17
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 13 | 9
Fall (Injury, poisoning and procedural complications) | 8 | 12
Hypoglycaemia (Metabolism and nutrition disorders) | 13 | 6
Septic shock (Infections and infestations) | 10 | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Hypertension (Vascular disorders) | 8 | 9
Coronary artery disease (Cardiac disorders) | 7 | 9
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Alanine aminotransferase increased (Investigations) | 7 | 8
Syncope (Nervous system disorders) | 6 | 9
Cardiac failure chronic (Cardiac disorders) | 7 | 7
Hip fracture (Injury, poisoning and procedural complications) | 12 | 2
Metabolic encephalopathy (Nervous system disorders) | 5 | 9
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 6
Diabetic nephropathy (Renal and urinary disorders) | 6 | 6
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Deep vein thrombosis (Vascular disorders) | 5 | 7
Hypertensive emergency (Vascular disorders) | 4 | 8
Acute left ventricular failure (Cardiac disorders) | 5 | 6
Myocardial infarction (Cardiac disorders) | 7 | 4
Osteomyelitis (Infections and infestations) | 5 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 6
Cerebrovascular accident (Nervous system disorders) | 7 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Left ventricular failure (Cardiac disorders) | 3 | 7
Clostridium difficile colitis (Infections and infestations) | 8 | 2
Urosepsis (Infections and infestations) | 6 | 4
Aspartate aminotransferase increased (Investigations) | 4 | 6
Ischaemic stroke (Nervous system disorders) | 8 | 2
Azotaemia (Renal and urinary disorders) | 4 | 6
Diabetic foot (Skin and subcutaneous tissue disorders) | 5 | 5
Angina unstable (Cardiac disorders) | 3 | 6
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 | 5
Transient ischaemic attack (Nervous system disorders) | 6 | 3
Hypertensive urgency (Vascular disorders) | 4 | 5
Pyelonephritis acute (Infections and infestations) | 3 | 5
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 6
Hypovolaemia (Metabolism and nutrition disorders) | 3 | 5
Encephalopathy (Nervous system disorders) | 3 | 5
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Hypotension (Vascular disorders) | 6 | 2
Atrial flutter (Cardiac disorders) | 2 | 5
Cardio-respiratory arrest (Cardiac disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 3 | 4
Multiple organ dysfunction syndrome (General disorders) | 4 | 3
Non-cardiac chest pain (General disorders) | 5 | 2
Gangrene (Infections and infestations) | 3 | 4
Gastroenteritis (Infections and infestations) | 3 | 4
Peritonitis (Infections and infestations) | 4 | 3
Pyelonephritis chronic (Infections and infestations) | 4 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4
Hypervolaemia (Metabolism and nutrition disorders) | 4 | 3
Mental status changes (Psychiatric disorders) | 2 | 5
Renal impairment (Renal and urinary disorders) | 3 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Blood loss anaemia (Blood and lymphatic system disorders) | 2 | 4
Bradycardia (Cardiac disorders) | 4 | 2
Cardiogenic shock (Cardiac disorders) | 2 | 4
Cardiorenal syndrome (Cardiac disorders) | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Asthenia (General disorders) | 1 | 5
Cholecystitis acute (Hepatobiliary disorders) | 3 | 3
Influenza (Infections and infestations) | 3 | 3
Pyelonephritis (Infections and infestations) | 4 | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hypertensive crisis (Vascular disorders) | 0 | 6
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 3
Pancreatitis acute (Gastrointestinal disorders) | 3 | 2
Device related infection (Infections and infestations) | 2 | 3
Diverticulitis (Infections and infestations) | 3 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 4
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 | 3
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 3 | 2
Urinary tract obstruction (Renal and urinary disorders) | 3 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 3
Angina pectoris (Cardiac disorders) | 1 | 3
Cardiopulmonary failure (Cardiac disorders) | 3 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 3 | 1
Gastritis (Gastrointestinal disorders) | 3 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Chest pain (General disorders) | 1 | 3
Generalised oedema (General disorders) | 2 | 2
Bronchitis (Infections and infestations) | 3 | 1
Cystitis (Infections and infestations) | 2 | 2
Device related sepsis (Infections and infestations) | 2 | 2
Peritonitis bacterial (Infections and infestations) | 2 | 2
Pneumonia bacterial (Infections and infestations) | 2 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Urinary tract infection bacterial (Infections and infestations) | 3 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 2
Hepatic enzyme increased (Investigations) | 1 | 3
Transaminases increased (Investigations) | 1 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Haemorrhagic stroke (Nervous system disorders) | 3 | 1
Seizure (Nervous system disorders) | 2 | 2
Depression (Psychiatric disorders) | 1 | 3
Renal tubular necrosis (Renal and urinary disorders) | 3 | 1
Aortic stenosis (Vascular disorders) | 2 | 2
Peripheral artery thrombosis (Vascular disorders) | 4 | 0
Peripheral ischaemia (Vascular disorders) | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Atrioventricular block (Cardiac disorders) | 1 | 2
Atrioventricular block complete (Cardiac disorders) | 1 | 2
Atrioventricular block second degree (Cardiac disorders) | 1 | 2
Coronary artery stenosis (Cardiac disorders) | 1 | 2
Pericardial effusion (Cardiac disorders) | 2 | 1
Pericarditis (Cardiac disorders) | 1 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 2
Hypothyroidism (Endocrine disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Catheter site haemorrhage (General disorders) | 1 | 2
Complication associated with device (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 1 | 2
Pyrexia (General disorders) | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 2
Abscess limb (Infections and infestations) | 2 | 1
Anal abscess (Infections and infestations) | 2 | 1
Appendicitis (Infections and infestations) | 0 | 3
Arteriovenous fistula site infection (Infections and infestations) | 1 | 2
Diabetic foot infection (Infections and infestations) | 2 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 2
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 3
Viral infection (Infections and infestations) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 2
Gout (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Device dislocation (Product Issues) | 0 | 3
Delirium (Psychiatric disorders) | 2 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 3
Glomerulonephritis (Renal and urinary disorders) | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 2
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 2
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
General physical health deterioration (General disorders) | 2 | 0
Sudden death (General disorders) | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 2
Liver injury (Hepatobiliary disorders) | 1 | 1
Kidney transplant rejection (Immune system disorders) | 0 | 2
Transplant rejection (Immune system disorders) | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 2
Clostridium difficile infection (Infections and infestations) | 2 | 0
Endocarditis (Infections and infestations) | 1 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 2
Escherichia sepsis (Infections and infestations) | 0 | 2
Intervertebral discitis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Pneumococcal sepsis (Infections and infestations) | 1 | 1
Pneumonia staphylococcal (Infections and infestations) | 2 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Arteriovenous fistula maturation failure (Injury, poisoning and procedural complications) | 2 | 0
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 2
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Blood potassium increased (Investigations) | 0 | 2
International normalised ratio increased (Investigations) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Obesity (Metabolism and nutrition disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2
Dementia (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 1
Uraemic encephalopathy (Nervous system disorders) | 2 | 0
Device occlusion (Product Issues) | 0 | 2
Cystitis haemorrhagic (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Arteriosclerosis (Vascular disorders) | 1 | 1
Hypovolaemic shock (Vascular disorders) | 2 | 0
Steal syndrome (Vascular disorders) | 1 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 1
Heart valve incompetence (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral valve calcification (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Pericarditis uraemic (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1
Tachycardia induced cardiomyopathy (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 1 | 0
Cataract diabetic (Eye disorders) | 1 | 0
Tractional retinal detachment (Eye disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyschezia (Gastrointestinal disorders) | 1 | 0
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hypothermia (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Treatment noncompliance (General disorders) | 0 | 1
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0
Gallbladder rupture (Hepatobiliary disorders) | 0 | 1
Granulomatous liver disease (Hepatobiliary disorders) | 0 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 1
Steatohepatitis (Hepatobiliary disorders) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abscess neck (Infections and infestations) | 0 | 1
Acute hepatitis C (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 0 | 1
Cardiac valve vegetation (Infections and infestations) | 0 | 1
Catheter bacteraemia (Infections and infestations) | 0 | 1
Catheter site cellulitis (Infections and infestations) | 1 | 0
Cryptosporidiosis infection (Infections and infestations) | 1 | 0
Cystitis bacterial (Infections and infestations) | 0 | 1
Cystitis klebsiella (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1
Endocarditis staphylococcal (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 0 | 1
Fournier's gangrene (Infections and infestations) | 0 | 1
Fungal peritonitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Gastritis viral (Infections and infestations) | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Intestinal sepsis (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0
Osteomyelitis bacterial (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Parotid abscess (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pneumonia escherichia (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Post procedural cellulitis (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Proteus infection (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyonephrosis (Infections and infestations) | 1 | 0
Renal graft infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Salmonella bacteraemia (Infections and infestations) | 1 | 0
Scarlet fever (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0
Serratia bacteraemia (Infections and infestations) | 0 | 1
Shunt infection (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Wound infection pseudomonas (Infections and infestations) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Device placement issue (Injury, poisoning and procedural complications) | 1 | 0
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood glucose fluctuation (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Electrocardiogram repolarisation abnormality (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy endocrine (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain stem stroke (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral artery thrombosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Diabetic coma (Nervous system disorders) | 1 | 0
Diabetic encephalopathy (Nervous system disorders) | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Lacunar stroke (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0
Thrombotic stroke (Nervous system disorders) | 0 | 1
VIth nerve disorder (Nervous system disorders) | 0 | 1
Vertigo CNS origin (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Anger (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Acute phosphate nephropathy (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 1 | 0
Glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Reflux nephropathy (Renal and urinary disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 1 | 0
Renal papillary necrosis (Renal and urinary disorders) | 1 | 0
Renal vascular thrombosis (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Capillaritis (Skin and subcutaneous tissue disorders) | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash scarlatiniform (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 0 | 1
Lymphorrhoea (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Subclavian vein stenosis (Vascular disorders) | 1 | 0
Vascular rupture (Vascular disorders) | 1 | 0
Vascular stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat (N=861) | Darbepoetin Alfa (N=862)
Hypertension (Vascular disorders) | 120 | 123
Urinary tract infection (Infections and infestations) | 93 | 113
Diarrhoea (Gastrointestinal disorders) | 117 | 76
Oedema peripheral (General disorders) | 84 | 85
Hyperkalaemia (Metabolism and nutrition disorders) | 71 | 78
Nausea (Gastrointestinal disorders) | 73 | 57
Fall (Injury, poisoning and procedural complications) | 64 | 53
Nasopharyngitis (Infections and infestations) | 53 | 61
Upper respiratory tract infection (Infections and infestations) | 55 | 44
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 | 48
Constipation (Gastrointestinal disorders) | 44 | 38
Bronchitis (Infections and infestations) | 44 | 32
Headache (Nervous system disorders) | 22 | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT02680574/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT02680574/SAP_001.pdf